CLINICAL TRIAL: NCT05577910
Title: Vectored Thermal Pulsation, Intense Pulsed Light, and Eyelid Warm Compress (VIEW) Therapies for Meibomian Gland Dysfunction- a Randomized, Assessor-masked, Active-controlled Clinical Trial
Brief Title: Vectored Thermal Pulsation, Intense Pulsed Light, and Eyelid Warm Compress Therapies for MGD
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Kelvin Kam-lung Chong, MD, Associate Professor, Department of Ophthalmology and Visual Sciences, CUHK, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HMRF-08190266
Record Dates: First submitted 2022-09-27; First posted 2022-10-13 (Actual); Last update posted 2025-02-19 (Actual); Status verified 2025-02

CONDITIONS: Meibomian Gland Dysfunction
Keywords: Meibomian Gland Dysfunction; Dry Eye Disease; Vectored Thermal Pulsation therapy; Intense Pulsed Light therapy
MeSH Terms: conditions — Meibomian Gland Dysfunction; Dry Eye Syndromes | interventions — Therapeutics; Ophthalmic Solutions; Hypromellose Derivatives

STUDY DESIGN:
Intervention Model Description: This is a prospective, randomized, assessor-masked, 3-arm (1:1:1), active-controlled trial of 360 subjects with meibomian gland dysfunction contributing one study eye. For subjects with both eyes eligible, the eye with the most meibomian gland dropout (meiboscore), fewest expressible meibomian glands, thinnest lipid layer, or lowest TFBUT values (in this order) will be selected as the study eye.
  Enrolled patients will be randomized into one of the following groups, 1 month after recruitment during the 15-month study period receiving bilateral treatment of:
  Group A: 1-session VTP at month 0
  Group B: 4-session IPL+MGX at month 0,1,2,3
  Group C: twice daily EW for 15 months
  Topical lubricating eye drops (Hypromellose, 3mg/ml) will be the monotherapy for all subjects.
Who Masked: Outcomes Assessor
Masking Description: Unmasked trial coordinators will ensure masking by reminding and accompanying each patient before and during visits. Treatment related complications will be evaluated by all participants in a standard datasheet regardless of group assignment. Follow-up investigators will be asked if they know each participant's group assignment at each visit and why.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (3):
- Group A (Experimental): One session VTP at month 0.
  Interventions: Device: Vectored thermal pulsation (VTP) therapy; Drug: Topical eye drops (Hypromellose, 3mg/ml)
- Group B (Experimental): Four sessions IPL+MGX at month 0,1,2,3.
  Interventions: Device: Intense pulsed light with meibomian gland expression (IPL+MGX) therapy; Drug: Topical eye drops (Hypromellose, 3mg/ml)
- Group C (Active Comparator): Twice daily EW for 15 months.
  Interventions: Behavioral: Eyelid Warm Compress Therapy (EW); Drug: Topical eye drops (Hypromellose, 3mg/ml)

INTERVENTIONS:
Device: Vectored thermal pulsation (VTP) therapy — VTP purchased from TearScience®️ is an automated thermal pulsation system that is designed to heat and simultaneously evacuate the meibomian gland contents. It is performed by the unmasked treating investigators as described by the equipment manufacturer. In brief, one to two drops of topical anesthesia are applied prior to the bilateral application of the activators. The inner portion of the activator applies a constant temperature of 42.5°C to the tarsal conjunctiva of upper and lower eyelids. Simultaneously, the outer portion of the activator applies directional, pulsatile pressure to the external eyelid surfaces (maximum 6 psi) for the 12-minute treatment cycle. Participants will receive one session of VTP treatment only (month 0).
  Arms: Group A
Device: Intense pulsed light with meibomian gland expression (IPL+MGX) therapy — IPL is delivered using the proprietary "dry eye mode" setting of the Lumenis®️ M22TM system per the Toyos protocol. Pulse intensity (11-14 J/cm2) is inversely related to the Fitzpatrick skin phototype of each participant and will be used for the same patient throughout the study. IPL will be delivered to four overlapping zones inferior to each eye and a fifth pulse applied temporally adjacent to the lateral canthus four times. Both eyelids are closed and sealed with IPL-Aid disposable eye shields. MGX is immediately performed on both upper and lower eyelids of each eye and pain will be minimized by topical anesthetic. Participants will receive four-session IPL and MGX treatment (month 0, 1, 2 ,3).
  Arms: Group B
Behavioral: Eyelid Warm Compress Therapy (EW) — EW using warm wet towel to each eye is performed twice daily for 10 mins. A treatment diary will be given for patients randomized to EW for daily recording which will be reviewed and recorded by the unmasked study coordinator at each study visit.
  Arms: Group C
Drug: Topical eye drops (Hypromellose, 3mg/ml) — All patients will be given one single topical lubricant (Hypromellose, 3mg/ml) to be used as frequently as needed from recruitment to study exit (total 16 months).

SUMMARY:
Meibomian gland dysfunction (MGD), closely associated with Dry Eye Disease (DED), is a chronic condition where terminal ducts are obstructed and/or glandular secretion changes. The efficacy of traditional treatment options, e.g. eyelid warm compress therapy (EW) is limited with low compliance. This study aims to (1)compare the efficacy and safety of two emerging alternatives- vectored thermal pulsation(VTP) or intense pulsed light and meibomian gland expression(IPL + MGX) with EW therapy; (2)identify factors predicting outcome.

This is a prospective, randomized, assessor-masked, active-controlled clinical study. 360 participants (360 study eyes) with mild-to-moderate MGD will be randomized by minimization into three arms equally, receiving either VTP by TearScience-LipiFlow® Thermal Pulsation System (month 0), IPL by Lumenis®️M22 with MGX (month 0, 1, 2, 3) or EW (twice daily). Lubricating eye drops (3% Hypromellose) will be provided for all subjects throughout the study period(15 months). Tear film breakup time will be assessed as primary outcome at month 6, 15. Serial measurements of MG, tear-film, DED-related parameters, intraocular pressure, compliance to EW, factors associated with outcomes and treatment-related complications will be conducted at baseline and each follow-up visit by masked observers at baseline and eight follow-up evaluation (month 0, 1, 2, 3, 4, 6, 9, 12, 15).

DETAILED DESCRIPTION:
Dry eye disease (DED) is an emerging, under-recognized and under-treated epidemic of the 21st century. It is one of the commonest reasons seeking eye consultation worldwide. Depending on the diagnostic criteria, geographic location and population concerned, prevalence of DED ranges from 30 to over 50% in the Asia Pacific regions compared to around 5-10% in the United States. Up to 90% of DED is closely associated with meibomian gland dysfunction (MGD), a chronic and progressive condition characterized by terminal duct obstruction, qualitative and/or quantitative changes in the glandular secretions (meibum) which causes tear instability by increasing tear evaporation and subsequently increased tear osmolarity, ocular surface inflammation, epithelial damage and ocular surface disease. Studies suggest that MGD affects between 5-20 % of Caucasians and over 60% of Asians populations.

Conventional treatments for MGD including self-administered eyelid hygiene, eyelid warm compress therapy (EW), artificial tears, including lipid-containing lubricants are limited in their efficacies for moderate to advanced disease. Prescription medications (topical steroids, topical and oral antibiotics, topical immunomodulatory agents e.g. cyclosporine and oral omega-3 essential fatty acids) have demonstrated efficacies in improving symptoms and signs of MGD; however side-effects including preservative-related adverse events, development of antibiotic resistance, cost, accessibility, off-label use, and the need for ongoing treatments often limit their long-term use.

Despite the described range of available options, management for MGDs is often considered unsatisfactory and frustrating by clinicians and patients. Compliance to long-term, home-based self-administered therapies is known to be suboptimal while practitioner-administered treatment including meibomian gland expression (MGX) provides transient relief.

Intense pulsed light (IPL) therapy is widely used in cosmetic dermatology as well as therapeutically for a wide range of skin conditions with favourable efficacy and tolerability. Concurrent MGD improvements were observed serendipitously in patients undergoing IPL for rosacea. With growing interest in combining IPL+MGX as practitioner-administered physical therapy for MGD, recent review and meta-analysis showed its effectiveness and safety while calling to investigate its effect beyond 6 months after the last IPL treatment.

Vectored thermal pulsation (VTP) is approved by FDA as another practitioner-administered physical therapy for MGD. The device covers both the cutaneous and mucosal surfaces of the eyelids; the rear portion of the device provides heat to the MG, and the front portion gives mechanical stimulation to the eyelid skin. It evacuates the MG of the upper and lower eyelids simultaneously with minimal discomfort while protecting the cornea, rendering the experience for patients generally favorable. Recent meta-analysis showed that a single 12-minute VTP was more efficacious than EW in treating MGD.

Knowledge gaps:

Level I evidence comparing efficacies between two promising practitioner-administered therapies VTP and multi-session IPL+MGX with standard self-administered twice-daily EW for MGD is currently lacking. The onset and offset of therapeutic effects, time course of multi-session IPL+MGX, single-session VTP or twice-daily EW on MGD up to 15-month post-treatment initiation or 12-month post last session of IPL have not been studied either in an RCT setting. These important gaps will be addressed in this application.

Primary Objective:

To compare the efficacy and safety of 1-session vectored thermal pulsation (VTP) or 4-session intense pulsed light and meibomian gland expression (IPL+MGX) with twice-daily eyelid warm compress (EW) therapy for meibomian gland dysfunction (MGD).

Secondary Objectives:

1. To compare the course of MGD among groups over 15 months (12-month after final IPL+MGX);
2. To identify factors predicting responses and compliance to therapies.

Hypotheses:

1. Both 1-session VTP and 4-session IPL+MGX are more efficacious than twice-daily EW in improving MGD;
2. MGD improves earlier after VTP;
3. MGD improvement lasts longer after 4-session IPL+MGX.

Study design:

This is a prospective, randomized, assessor-masked, 3-arm (1:1:1), active-controlled trial of 360 subjects with meibomian gland dysfunction contributing one study eye. For subjects with both eyes eligible, the eye with the fewest quality of expressed meibum, thinnest lipid layer, or the lowest TFBUT values (in this order) will be selected as the study eye.

A total of 360 patients with symptomatic MGD will be recruited from the participating hospitals coordinated by the Chinese University of Hong Kong (CUHK) Research Clinic, the CUHK Eye Centre (CUHKEC), Department of Ophthalmology and Visual Science, Faculty of Medicine, The CUHK.

Randomization will be carried out by a computer-generated minimization program. Minimization is a dynamic process to reduce the imbalance between trial arms with respect to a range of predefined prognostic variables, and a randomization schedule is therefore not drawn up in advance. A form describing the baseline characteristics of each subject according to these minimization criteria: gender, age, and quality of expressed meibum from the study eye. Treatment allocation will be sent to the unmasked trial coordinator for arrangement at baseline (month 0).

Enrolled patients will be randomized into one of the following groups, 1 month after recruitment during the 15-month study period receiving bilateral treatment of:

Group A: 1-session VTP at month 0; Group B: 4-session IPL+MGX at month 0,1,2,3; Group C: twice daily EW for 15 months.

All patients will be given one single topical lubricant (Hypromellose, 3mg/ml) to be used as frequently as needed from recruitment to study exit (total 16 months).

IPL or VTP is given by unmasked treating investigators not involved in data collection. Follow-up investigators collecting the data are masked to participants' treatment assignment. This information can be disclosed upon request after the completion of the study. Unmasked trial coordinators will ensure masking by reminding and accompanying each patient before and during visit. Treatment-related complications will be evaluated by all participants in a standard datasheet regardless of group assignment. Follow-up investigators will be asked if they know each participant's group assignment at each visit and why.

Tear film breakup time will be assessed as the primary outcome (month 6 and 15). Serial measurements of MG, tear-film, DED-related parameters, intraocular pressure, compliance to EW, factors associated with outcomes, and treatment-related complications will be conducted by masked investigators at baseline and eight follow-up evaluations (month 0, 1, 2, 3, 4, 6, 9, 12, 15).

ELIGIBILITY:
Inclusion Criteria:

1. ≥18 years of age with no upper age limit;
2. Agree to attend follow-up visits and comply to treatment regimen;
3. Symptomatic dry eye TFBUT (average of 3 times) ≤ 5 seconds and OSDI ≥ 13;
4. Mild to moderate (level 3-4) MGD on at least one eye;
5. Fitzpatrick skin type 1-4.

Exclusion Criteria:

1. Contact lens wear 3 months before or during the study period;
2. Use of topical (including anti-glaucomatous, cyclosporin, antibiotics) or systemic medication known to affect (worsen or improve) MGD 3 months before or during the study period;
3. Major systemic (e.g. Sjogren's syndrome), dermatologic (e.g. Rosacea) known to affect MGD or ocular conditions (including thyroid eye disease, recurrent conjunctivitis, ocular allergies);
4. Ocular procedures (excluding uncomplicated cataract operation) 3 months before and any ocular procedure during the study period;
5. History of vision correction surgery or plan to undergo the procedure during the study period;
6. Dermatological treatment (including chemical peeling, laser, IPL or energy device in the periocular and facial region) 6 months before or during the study period;
7. Contraindications to IPL therapy (including recent sun-burn, photosensitivity, active or pigmented skin lesions, cancer, implants, tattoos, semi-permanent makeup in the periocular area);
8. Contraindications to VTP therapy (ocular surgery, ocular injury, ocular herpes of eye or eyelid, and ocular inflammation 3 months before the study; active ocular infection, etc.)
9. Women who are pregnant, nursing, planning pregnancy, or of childbearing potential not using a reliable method of contraception.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 360 (Estimated)
Dates: Start 2022-10-08 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Change from baseline Tear film breakup time (TFBUT) at 6 months | 6 months
  Sodium fluorescein will be instilled in both eyes of the subject. A follow-up investigator will do the examination by slit lamp. Tear film breakup time (TFBUT) is the time to initial breakup of the tear film after a blink is measured three times and taken average.
Change from baseline Tear film breakup time (TFBUT) at 15 months | 15 months
  Sodium fluorescein will be instilled in both eyes of the subject. A follow-up investigator will do the examination by slit lamp. Tear film breakup time (TFBUT) is the time to initial breakup of the tear film after a blink is measured three times and taken average.

SECONDARY OUTCOMES:
Change in Ocular Surface Disease Index (OSDI) | 15 months
  The 12-item symptom frequency-based questionnaire Ocular Surface Disease Index (OSDI) is self-administered by patients at each study visit for assessment of dry eye disease (DED) related symptoms and its severity. Final OSDI score is calculated by dividing the product of the total sum of score and 25 by the total number of answered questions, with a range from 0 to 100 (normal: 0-12, mild dry eye disease: 13-22, moderate dry eye disease: 23-32, severe dry eye disease: >33).
Change in Standard Patient Evaluation of Eye Dryness (SPEED) | 15 months
  The Standard Patient Evaluation of Eye Dryness (SPEED) questionnaire is self-administered by patients at each study visit for monitoring dry eye symptoms progression throughout the study. Final SPEED score is calculated by summating the score of all answered questions, with a range from 0 to 28 (mild dry eye symptoms: 0-4, moderate dry eye symptoms: 5-7, severe dry eye symptoms: >8).
Change in symptom Assessment iN Dry Eye (SANDE) | 15 months
  The 2-item frequency- and severity-based visual analog scale Symptom Assessment iN Dry Eye (SANDE) questionnaire is self-administered by patients at each study visit to evaluate the frequency and severity of dry eye symptoms. Final SANDE score is calculated by obtaining the square root of the product of the frequency of symptoms score and the severity of symptoms score, with a range from 0 (minimal degree of dry eye symptoms) to 100 (maximal degree of dry eye symptoms)
Change in ocular comfort index (OCI) | 15 months
  The Ocular Comfort Index (OCI) questionnaire is self-administered by patients at each study visit to evaluate the topical treatment outcome of dry eye symptoms. The final OCI score will be linearly rescaled which ranges from 0 (minimal degree of dry eye symptoms) to 100 (maximal degree of dry eye symptoms).
Change in dry eye questionnaire (DEQ-5) | 15 months
  The Dry Eye Questionnaire (DEQ-5) is self-administered by patients at each study visit for assessment of the frequency and intensity of dry eye symptoms. The final DEQ-5 score is calculated by summating the score of all answered questions, with a range from 0 to 22. A score greater or equal to 6 is considered positive for dry eye symptoms.
Change in tear film breakup time (TFBUT) | 15 months
  Sodium fluorescein will be instilled in both eyes of the subject. A follow-up investigator will do the examination by slit lamp. Tear film breakup time (TFBUT) is the time to initial breakup of the tear film after a blink is measured three times and taken average.
Change in non-invasive keratograph break-up time (NIKBUT) | 15 months
  Non-invasive keratograph break-up time (NIKBUT) is measured using automated detection of the first break-up by Keratograph 5M (OCULUS, Wetzlar, Germany), while the subject maintains fixation and is requested to refrain from blinking. Three break-up time readings are averaged in each case for both eyes.
Change in bulbar conjunctival hyperaemia | 15 months
  Bulbar conjunctival hyperaemia is evaluated by Keratograph 5M (OCULUS, Wetzlar, Germany) according to the proprietary JENVIS grading scale from 0 to 4.
Change in lower tear meniscus height (TMH) | 15 months
  The lower tear meniscus height (TMH) is assessed using high magnification pre-calibrated digital imaging by Keratograph 5M (OCULUS, Wetzlar, Germany), and three measurement points (nasal and temporal limbus, pupil center) of the lower meniscus are averaged.
Change in lipid layer thickness (LLT) | 15 months
  Lipid layer thickness (LLT) of the tear film as determined with LipiView II (TearScience, Morrisville, NC). Minimum, Maximum and Average thickness in nm will be measured.
Change in tear interferometric fringe pattern | 15 months
  Tear interferometric fringe pattern is graded according to the modified Guillon-Keeler system with LipiView II (TearScience, Morrisville, NC). It will be graded according to the modified Guillon-Keeler system: grade 1, open meshwork; grade 2, closed meshwork; grade 3, wave or flow; grade 4, amorphous; grade 5, colored fringes; grade 0, non-continuous layer (non-visible or abnormal colored fringes).
Change in meiboscore | 15 months
  The meiboscore grading scale uses a 0 to 3 grading scale by LipiView II (TearScience, Morrisville, NC) infrared meibography on both superior and inferior eyelids, with a grade of 0 representing no meibomian gland atrophy, with grades of 1, 2, and 3 representing 1% to 33%, 34% to 66%, and ≥67% of glands lost, respectively.
Change in meibograde | 15 months
  Meibograde is evaluating gland distortion, gland shortening, and gland dropout by LipiView II (TearScience, Morrisville, NC) infrared meibography on both superior and inferior eyelids. Each of these characteristics is graded from 0-3, like the meiboscore, and then they are summed to give a total score of 0-9 per eyelid.
Change in partial blinking rate | 15 months
  Partial blinking rate is reported as the percentage of incomplete blinks, which recorded by LipiView II (TearScience, Morrisville, NC).
Change in schirmer's test (ST) | 15 months
  Schirmer's test (ST) will be performed by standard filter paper strips without anesthesia for 5 mins in both eyes at the same time. The wetting length by tears in each strip is recorded. The strips will be collected in sterile centrifuge tubes respectively for laboratory tests.
Change in Lid margin and eyelash abnormalities | 15 months
  Lid margin and eyelash abnormalities will be accessed by a slit lamp, including lid margin thickening, rounding, notching, foaming, telangiectasia, meibomian gland capping, staphylococcal lash crusting, seborrheic lash crusting, Demodex lash cylindrical collarettes, madarosis, poliosis, and trichiasis.
  All items will be graded based on a four-point scale: grade 0, absent; grade 1, mild; grade 2, moderate; grade 3, severe.
Change in corneal and conjunctival staining score | 15 months
  Corneal and conjunctival damage is evaluated by corneal and conjunctival staining scores according to the Oxford grading system (six-point scale). Fluorescein sodium will be Instilled in both eyes. The staining of the eyes will be examined by follow-up investigators with a slit lamp under cobalt blue light.
  Scores range from 0-5 ( absent to severe).
Change in lid wiper epitheliopathy (LWE) | 15 months
  Lid wiper epitheliopathy (LWE) is evaluated relative to Korb's grading. Only the superior eyelid will be examined on the linear area of staining and severity of staining.
  The linear area of staining is graded on a three-point scale (grade 0, <2 mm; grade 1, 2-4 mm; grade 2, 5-9 mm; grade 3, ≥10 mm).
  The severity of staining is graded on a four-point scale (grade 0, none; grade 1, slight; grade 2, mild; grade 3, moderate; grade 4, severe).
  The total grade was the sum of the grading score of the linear area of staining and severity of staining.
Change in expressibility of meibomian glands in the meibomian glands yielding liquid secretion (MGYLS) (the inferior eyelid) | 15 months
  Expressibility of the inferior eyelid meibomian glands is assessed with the Meibomian Gland Evaluator (TearScience, North Carolina, USA) applied just inferior to the nasal, central, and temporal aspects of the inferior eyelid margin.
  The meibomian glands yielding liquid secretion (MGYLS) is the total number of glands which yielding lipid secretions at the nasal, central, and temporal aspects of the eyelid margin (5 glands each part).
Change in expressibility of meibomian glands in proportion of meibomian orifices yielding lipid secretions (the inferior eyelid)) | 15 months
  Expressibility of the inferior eyelid meibomian glands is assessed with the Meibomian Gland Evaluator (TearScience, North Carolina, USA) applied just inferior to the nasal, central, and temporal aspects of the inferior eyelid margin.
  The proportion of meibomian orifices yielding lipid secretions is graded on a five-point scale: 0, more than 75% (4-5 glands); 1, 50% to 75% (3 glands); 2, 25% to 50% (2 glands); 3, less than 25% (1 gland); 4, none (0 gland).
Change in quality of expressed meibum | 15 months
  Each gland in each area is assessed for expressibility and graded according to a 4-point scale (grade 0, no secretion; grade 1, inspissated/ toothpaste-like expression; grade 2, cloudy fluid secretion; and grade 3, clear fluid/normal secretion). The sum scores of 15 glands will be between 0 and 45.

OTHER OUTCOMES:
Change in visual acuity | 15 months
  Visual acuity is examined by standard visual acuity chart as safety outcome measures.
Levels in procedure-related pain (VAS) | 3 months
  Procedure-related pain (VAS) is graded on a ten-point score (from no pain, moderate pain, to worst pain) as safety outcome measures.
Change in intraocular pressure | 15 months
  The intraocular pressure, the fluid pressure of the eye, is assessed by a non-contact tonometer as the safety outcome measure.
Change in lens opacity | 15 months
  Lens opacity is graded by the slip lamp according to the Lens Opacities Classification System (LOCS II) as a safety outcome measure. There are 4 standards for nuclear grading (grade 0/1/2/3), 5 standards for cortical grading (0/TR/1/2/3/4/5), and 4 standards for posterior grading (0/1/2/3/4).
Change in anterior chamber activities | 15 months
  Anterior chamber activities are graded by the Standardization of Uveitis Nomenclature (SUN) grading system: 1) cells (0/0.5+/1+/2+/3+/4+); 2) flare (0/1+/2+/3+/4+).
Number of participants with iris defect and transillumination | 15 months
  Iris defect and transillumination are assessed by 2-point scale as safety outcome measure. (0: no; 1: absent).
Number of participants with abnormalities of fundus | 15 months
  Both of the subject's eyes will be dilated. The fundus examination is performed by a follow-up investigator, and abnormalities of fundus will be recorded. The number of participants with the situation will be counted.
Number of participants with loss of lashes and eyebrows | 15 months
  Loss of lashes and eyebrows are assessed by 2-point scale as safety outcome measure. (0: no; 1: absent). The number of participants with the situation will be counted.
Number of participants with facial redness | 15 months
  Facial redness is assessed by 2-point scale as safety outcome measure. (0: no; 1: absent). The number of participants with the situation will be counted.
Number of participants with facial swelling | 15 months
  Facial swelling is graded by 2-point scale as safety outcome measure. (0: no; 1: absent). The number of participants with the situation will be counted.
Number of participants with facial bruises | 15 months
  Facial bruises are graded by 2-point scale as safety outcome measure. (0: no; 1: absent). The number of participants with the situation will be counted.
Number of participants with facial pigmentation | 15 months
  Facial pigmentation is graded by 2-point scale as safety outcome measure. (0: no; 1: absent). The number of participants with the situation will be counted.
Change of α-diversity in ocular surface microbiome | 15 months
  Each eye will be sampled by a sterile, polyester swab on the inferior fornix of the conjunctiva. The swabs will be placed in 2 mL microcentrifuge tubes at 4 °C. Extraction will be performed by laboratory staff, then the sample will be transferred to -80 °C laboratory freezer for long-term storage before further gene expression tests. After genomic DNA extraction from conjunctival swab samples for 16S rRNA sequencing, the resulting amplicons will be filtered, clustered into operational taxonomic units (OTUs) and taxonomically classified using reference databases. The α-diversity will be calculated and reported as ordination plots.
Change of β-diversity in ocular surface microbiome | 15 months
  Each eye will be sampled by a sterile, polyester swab on the inferior fornix of the conjunctiva. The swabs will be placed in 2 mL microcentrifuge tubes at 4 °C. Extraction will be performed by laboratory staff, then the sample will be transferred to -80 °C laboratory freezer for long-term storage before further gene expression tests. After genomic DNA extraction from conjunctival swab samples for 16S rRNA sequencing, the resulting amplicons will be filtered, clustered into operational taxonomic units (OTUs) and taxonomically classified using reference databases. The β-diversity will be calculated and reported as ordination plots.
Gene expression profiles | Baseline
  Subjects' blood specimens will be collected at the baseline visit and pre-treated for further laboratory tests. After genomic DNA extraction from venous blood, Single-nucleotide polymorphism (SNP) will be selected, sequenced and compared between treatment groups for pharmacogenomic analyses.

CONTACTS AND LOCATIONS:
Overall Officials: Kelvin KL Chong, MBChB, Principal Investigator — The Department of Ophthalmology & Visual Sciences, the Chinese University of Hong Kong
Locations (4):
- Hong Kong (4):
  - Hong Kong Eye Hospital, Kowloon, Hong Kong
  - The Chinese University of Hong Kong Eye Centre (CUHKEC), Kowloon
  - The CUHK Medical Centre (CUHKMC), Shatin
  - Prince of Wales Hospital, Shatin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Nelson JD, Craig JP, Akpek EK, Azar DT, Belmonte C, Bron AJ, Clayton JA, Dogru M, Dua HS, Foulks GN, Gomes JAP, Hammitt KM, Holopainen J, Jones L, Joo CK, Liu Z, Nichols JJ, Nichols KK, Novack GD, Sangwan V, Stapleton F, Tomlinson A, Tsubota K, Willcox MDP, Wolffsohn JS, Sullivan DA. TFOS DEWS II Introduction. Ocul Surf. 2017 Jul;15(3):269-275. doi: 10.1016/j.jtos.2017.05.005. Epub 2017 Jul 20. No abstract available. PMID 28736334
- [Background] Schein OD, Munoz B, Tielsch JM, Bandeen-Roche K, West S. Prevalence of dry eye among the elderly. Am J Ophthalmol. 1997 Dec;124(6):723-8. doi: 10.1016/s0002-9394(14)71688-5. PMID 9402817
- [Background] Chan TCY, Chow SSW, Wan KHN, Yuen HKL. Update on the association between dry eye disease and meibomian gland dysfunction. Hong Kong Med J. 2019 Feb;25(1):38-47. doi: 10.12809/hkmj187331. Epub 2019 Jan 31. PMID 30713149
- [Background] Schaumberg DA, Nichols JJ, Papas EB, Tong L, Uchino M, Nichols KK. The international workshop on meibomian gland dysfunction: report of the subcommittee on the epidemiology of, and associated risk factors for, MGD. Invest Ophthalmol Vis Sci. 2011 Mar 30;52(4):1994-2005. doi: 10.1167/iovs.10-6997e. Print 2011 Mar. No abstract available. PMID 21450917
- [Background] Nelson JD, Shimazaki J, Benitez-del-Castillo JM, Craig JP, McCulley JP, Den S, Foulks GN. The international workshop on meibomian gland dysfunction: report of the definition and classification subcommittee. Invest Ophthalmol Vis Sci. 2011 Mar 30;52(4):1930-7. doi: 10.1167/iovs.10-6997b. Print 2011 Mar. No abstract available. PMID 21450914
- [Background] Thode AR, Latkany RA. Current and Emerging Therapeutic Strategies for the Treatment of Meibomian Gland Dysfunction (MGD). Drugs. 2015 Jul;75(11):1177-85. doi: 10.1007/s40265-015-0432-8. PMID 26130187
- [Background] Wladis EJ, Bradley EA, Bilyk JR, Yen MT, Mawn LA. Oral Antibiotics for Meibomian Gland-Related Ocular Surface Disease: A Report by the American Academy of Ophthalmology. Ophthalmology. 2016 Mar;123(3):492-6. doi: 10.1016/j.ophtha.2015.10.062. Epub 2015 Dec 23. PMID 26707417
- [Background] Dry Eye Assessment and Management Study Research Group; Asbell PA, Maguire MG, Pistilli M, Ying GS, Szczotka-Flynn LB, Hardten DR, Lin MC, Shtein RM. n-3 Fatty Acid Supplementation for the Treatment of Dry Eye Disease. N Engl J Med. 2018 May 3;378(18):1681-1690. doi: 10.1056/NEJMoa1709691. Epub 2018 Apr 13. PMID 29652551
- [Background] Lam PY, Shih KC, Fong PY, Chan TCY, Ng AL, Jhanji V, Tong L. A Review on Evidence-Based Treatments for Meibomian Gland Dysfunction. Eye Contact Lens. 2020 Jan;46(1):3-16. doi: 10.1097/ICL.0000000000000680. PMID 31834043
- [Background] Foulks GN, Nichols KK, Bron AJ, Holland EJ, McDonald MB, Nelson JD. Improving awareness, identification, and management of meibomian gland dysfunction. Ophthalmology. 2012 Oct;119(10 Suppl):S1-12. doi: 10.1016/j.ophtha.2012.06.064. PMID 23034341
- [Background] Sabeti S, Kheirkhah A, Yin J, Dana R. Management of meibomian gland dysfunction: a review. Surv Ophthalmol. 2020 Mar-Apr;65(2):205-217. doi: 10.1016/j.survophthal.2019.08.007. Epub 2019 Sep 5. PMID 31494111
- [Background] Aketa N, Shinzawa M, Kawashima M, Dogru M, Okamoto S, Tsubota K, Shimazaki J. Efficacy of Plate Expression of Meibum on Tear Function and Ocular Surface Findings in Meibomian Gland Disease. Eye Contact Lens. 2019 Jan;45(1):19-22. doi: 10.1097/ICL.0000000000000535. PMID 30252688
- [Background] Toyos R, McGill W, Briscoe D. Intense pulsed light treatment for dry eye disease due to meibomian gland dysfunction; a 3-year retrospective study. Photomed Laser Surg. 2015 Jan;33(1):41-6. doi: 10.1089/pho.2014.3819. PMID 25594770
- [Background] Wladis EJ, Aakalu VK, Foster JA, Freitag SK, Sobel RK, Tao JP, Yen MT. Intense Pulsed Light for Meibomian Gland Disease: A Report by the American Academy of Ophthalmology. Ophthalmology. 2020 Sep;127(9):1227-1233. doi: 10.1016/j.ophtha.2020.03.009. Epub 2020 Apr 21. PMID 32327256
- [Background] Tashbayev B, Yazdani M, Arita R, Fineide F, Utheim TP. Intense pulsed light treatment in meibomian gland dysfunction: A concise review. Ocul Surf. 2020 Oct;18(4):583-594. doi: 10.1016/j.jtos.2020.06.002. Epub 2020 Jul 3. PMID 32629039
- [Background] Leng X, Shi M, Liu X, Cui J, Sun H, Lu X. Intense pulsed light for meibomian gland dysfunction: a systematic review and meta-analysis. Graefes Arch Clin Exp Ophthalmol. 2021 Jan;259(1):1-10. doi: 10.1007/s00417-020-04834-1. Epub 2020 Jul 28. PMID 32725403
- [Background] Pang SP, Chen YT, Tam KW, Lin IC, Loh EW. Efficacy of Vectored Thermal Pulsation and Warm Compress Treatments in Meibomian Gland Dysfunction: A Meta-Analysis of Randomized Controlled Trials. Cornea. 2019 Jun;38(6):690-697. doi: 10.1097/ICO.0000000000001907. PMID 30844843
- [Background] Sung J, Wang MTM, Lee SH, Cheung IMY, Ismail S, Sherwin T, Craig JP. Randomized double-masked trial of eyelid cleansing treatments for blepharitis. Ocul Surf. 2018 Jan;16(1):77-83. doi: 10.1016/j.jtos.2017.10.005. Epub 2017 Nov 8. PMID 29128682
- [Background] Foulks GN, Bron AJ. Meibomian gland dysfunction: a clinical scheme for description, diagnosis, classification, and grading. Ocul Surf. 2003 Jul;1(3):107-26. doi: 10.1016/s1542-0124(12)70139-8. PMID 17075643
- [Background] Bron AJ, Benjamin L, Snibson GR. Meibomian gland disease. Classification and grading of lid changes. Eye (Lond). 1991;5 ( Pt 4):395-411. doi: 10.1038/eye.1991.65. PMID 1743355
- [Background] Korb DR, Greiner JV, Herman JP, Hebert E, Finnemore VM, Exford JM, Glonek T, Olson MC. Lid-wiper epitheliopathy and dry-eye symptoms in contact lens wearers. CLAO J. 2002 Oct;28(4):211-6. doi: 10.1097/01.ICL.0000029344.37847.5A. PMID 12394549
- [Background] Guillon M, Maissa C. Assessment of upper and lower lid margin with lissamine green. Optom Vis Sci. 2008;84.
- [Background] Yamamoto Y, Shiraishi A, Sakane Y, Ohta K, Yamaguchi M, Ohashi Y. Involvement of Eyelid Pressure in Lid-Wiper Epitheliopathy. Curr Eye Res. 2016;41(2):171-8. doi: 10.3109/02713683.2015.1009636. Epub 2015 Mar 24. PMID 25803436
- [Background] Tomlinson A, Bron AJ, Korb DR, Amano S, Paugh JR, Pearce EI, Yee R, Yokoi N, Arita R, Dogru M. The international workshop on meibomian gland dysfunction: report of the diagnosis subcommittee. Invest Ophthalmol Vis Sci. 2011 Mar 30;52(4):2006-49. doi: 10.1167/iovs.10-6997f. Print 2011 Mar. No abstract available. PMID 21450918
- [Background] Korb DR, Blackie CA. Meibomian gland diagnostic expressibility: correlation with dry eye symptoms and gland location. Cornea. 2008 Dec;27(10):1142-7. doi: 10.1097/ICO.0b013e3181814cff. PMID 19034129